CLINICAL TRIAL: NCT05164497
Title: The Effect of Deliberate Practice Training of Graduate Students in General Psychotherapeutic Skills Compared to Theoretical Teaching: the Randomized Controlled TRIPS Trial
Brief Title: Training of Graduate Students in General Psychotherapeutic Skills (TRIPS)
Acronym: TRIPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Ole Karkov Østergård, Assistant Professor, PhD, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 201891619
Record Dates: First submitted 2021-11-10; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Deliberate Practice Training of Psychotherapeutic Skills; Theoretical Teaching of Psychotherapeutic Skills
Keywords: Psychotherapy training; Deliberate practice; Psychology students

STUDY DESIGN:
Intervention Model Description: Students will be individually randomized within each study site using a random number generator with a 1:1 allocation ratio, determining the order in which the experimental and control condition will be delivered. Half of the students will first receive the experimental condition, followed by the control condition, while the other half will receive the conditions in the reverse order. By the end of the course, all students will have received the same teaching and training, in reverse order. Main outcome analyses will be performed before the crossover (reflecting true randomization).
Who Masked: Outcomes Assessor
Masking Description: The blinding of raters will be ensured for the primary performance-based outcome (i.e., Facilitative Interpersonal Skills) by assigning the video-recorded responses randomly to the raters and concealing the group allocation (experimental vs. control) and time of measurement (week 0, 5, or 10). Furthermore, analyses of outcomes and the conclusion regarding hypotheses 1 and 2 will be performed blinded to allocation (i.e., results in favor of condition X or Y).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deliberate practice training (Experimental): The experimental condition consists of deliberate practice training of non-specific psychotherapy skills using role-play and Theravue, an online skill-building system with therapy videos.
  Interventions: Other: Deliberate practice training
- Theoretical teaching (Active Comparator): The control condition will consist of theoretical teaching of non-specific psychotherapy skills.
  Interventions: Other: Theoretical teaching

INTERVENTIONS:
Other: Deliberate practice training — The experimental condition consists of five weeks of deliberate practice training of non-specific psychotherapy skills organized as (1) classroom training and (2) homework. The classroom training consists of 15 hours (5 days x 3 hours) of deliberate practice training. Each day will be organized around a theme: (a) Empathy, (b) establishing the therapeutic alliance, (c) working with alliance ruptures, (d) formulation of an interpersonal focus, and (e) clinical expertise - a synthesis. The training will include theoretical introductions, students defining individual training goals, model responses of good psychotherapeutic skills, and student role-play. Regarding homework, after each of the five classes, the students will use Theravue to watch and respond to three therapy videos related to the theme of the previous class. The students have to deliver at least two new responses to each video informed by feedback from teachers and peers and a checklist describing a "good response."
  Arms: Deliberate practice training
Other: Theoretical teaching — The control condition will consist of five weeks of theoretical teaching of non-specific psychotherapy skills performed as (1) classroom teaching and (2) homework. Regarding classroom teaching, the 15 hours (5 days x 3 hours) of teaching will be organized around the same five themes as the experimental condition (see points a-d above). The class will consist of the teacher's presentation of theory and research findings, videos with master therapists defining core concepts, and group discussions of literature. Regarding homework, the participants will read literature and use a restricted version of Theravue to complete home assignments where they record their answers to three theoretical questions related to the theme of the preceding classroom teaching.
  Arms: Theoretical teaching

SUMMARY:
In this study, a deliberate practice-based approach to therapist training will be compared to theoretical teaching. The main hypothesis is that deliberate practice training will result in a larger improvement in students' observer-rated interpersonal skills. About 200 graduate students from two Danish universities will be randomized into two groups, a) deliberate practice training of non-specific psychotherapeutic skills using role-play and Theravue, an online skill-building system with therapy videos; or b) theoretical teaching. Each condition consists of 15 hours of classroom participation and homework. The study has the potential to transform the training of psychotherapy skills.

DETAILED DESCRIPTION:
Background: Psychology students at universities in Denmark and worldwide only receive little clinical training, even though such training is crucial to psychologists' job performance after graduation. Training non-specific psychotherapeutic skills, such as being empathic and facilitating the therapeutic alliance, is critical since these skills are related to psychotherapy outcomes. In this study, a deliberate practice approach to training will be compared to theoretical teaching.

Hypothesis: The first and main hypothesis is that the students' observer-rated Facilitative Interpersonal Skills (FIS) will improve significantly more after deliberate practice training compared to theoretical teaching. The second hypothesis is that students' self-reported Facilitative Interpersonal Skills (FIS-SR), self-efficacy, and empathy will increase significantly more after training compared to theoretical teaching. The third hypothesis is that students reporting higher baseline levels of self-affiliation, attachment security, external feedback propensity, and self-efficacy will have a larger increase in FIS after the training program. The fourth hypothesis is that the amount of deliberate practice will predict improvement in FIS at post-training, whereas the students' sociodemographic characteristics, previous experience with psychotherapy, and preferred psychotherapy approach will not be associated with improvement in FIS.

Methods: One hundred ninety-eight graduate students from the Universities of Copenhagen and Aalborg University will be randomized into two groups, a) deliberate practice training of non-specific skills using role-play and Theravue, or b) theoretical teaching. Group a will first receive the experimental condition (deliberate practice), followed by the control condition, while group b will receive the conditions in reverse order. Each condition consists of 15 hours of classroom participation and homework. The primary outcome is Facilitative Interpersonal Skills - Observer. Secondary outcomes include the Facilitative Interpersonal Skills-Self-Report, the Counselor Activity Self-Efficacy Scales, and the Interpersonal Reactivity Index. Outcomes will be measured at baseline (week 0), after the first condition (week 5; before the crossover, reflecting true randomization), and after both conditions (week 10). Main outcome analyses will be performed at week 5.

To test deliberate practice as a predictor of FIS improvement, the amount of deliberate practice activity is measured on a self-report questionnaire developed for this study and tracked on Theravue as a) the total time spent on watching and responding to therapy videos and b) the average number of attempts to improve the response to each therapy video. The Structural Analysis of Social Behavior Intrex questionnaire (SASB; Benjamin, 2000), the Social Skills Inventory (SSI; Riggio, 1989), the Experiences in Close Relationships Scale (ECR; Brennan et al., 1998), and the Internal and External Feedback Propensity Scales (IEFPS; Herold et al., 1996) will be measured at week 0 and explored as possible between-condition moderators of the outcome. The Group Climate Questionnaire-Short Form (GCQ-S; MacKenzie, 1983) will be used to measure the collaboration in the student groups, where approximately five students work together throughout the study period, performing role-plays and giving peer feedback in the experimental condition, and discussing theory in the control condition. The observer-rated DP Coach Competency Scale (DPCCS; Rousmaniere, 2020) will be used to evaluate adherence and quality of the deliberate practice training. Stig Bernt Poulsen, University of Copenhagen, and Ole Karkov Østergård, Aalborg University, are co-principal investigators.

Discussion: The study can potentially transform the training of psychotherapy, not only for psychology students but also for psychologists in general. Furthermore, the results of the study can be transferred to the training of other clinical skills.

Ethics: Ethical approval has been obtained from the Institutional Ethical Review Board, Department of Psychology, University of Copenhagen, and Aalborg University. Before signing up for the course, the students will be informed about the course and the research embedded herein. Informed consent will be obtained from students agreeing to participate in the study. Course participants can decline to participate in the study without negative consequences for their course participation.

ELIGIBILITY:
Inclusion Criteria:

* Graduate psychology students attending a 30-hour elective course in clinical psychology called "Deliberate practice training of general psychotherapeutic skills" at two universities in Denmark (i.e., Department of Communication and Psychology at Aalborg University and the Department of Psychology at the University of Copenhagen).
* All participants hold a Bachelor of Science in psychology.
* Signed informed consent.

Exclusion Criteria:

* Course participants who are declining to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Facilitative Interpersonal Skills - Observer (FIS; Anderson & Patterson, 2013) | Three different sets, each consisting of three FIS videos, will be presented to each student three times in randomized order: at baseline (week 0), after the first condition (week 5), and after the second condition (week 10)
  FIS measures relationship skills exhibited in psychotherapy. The therapists are asked to respond as helpfully as possible to video clips simulating challenging therapy situations. FIS has eight dimensions: (1) verbal fluency; (2) hope and positive expectations; (3) persuasiveness; (4) emotional expression; (5) warmth, acceptance, and understanding; (6) empathy; (7) alliance-bond capacity; and (8) alliance rupture-repair responsiveness. The items are rated on a 5-point Likert scale from 1 = skill deficit to 5 = optimal presence of skill.

SECONDARY OUTCOMES:
Change in Facilitative Interpersonal Skills-Self-Report (FIS-SR, Anderson, et al., 2020) | Immediately after replying to the FIS videos at week 0, week 5, and week 10
  FIS-SR measures self-evaluated relationship skills. Following participation in the FIS task, participants rate their performance on the eight FIS dimensions mentioned above. Participants rate the extent to which they believe that their FIS responses were verbally fluent, communicated hope and positive expectations, etc., on a 5-point Likert scale ranging from 1 = strongly disagree to 5 = strongly agree.
Change in Counselor Activity Self-Efficacy Scales (CASES; Lent et al., 2003) | Week 0, week 5, and week 10
  The CASES measure therapist's experience of self-efficacy within various domains. The present study uses the 15 items measuring Helping Skill Self-Efficacy, and the 10 items measuring Session Management Self-Efficacy. Each item is rated on a 10-point Likert scale ranging from 0 = no confidence to 9 = complete confidence.
Change in Interpersonal Reactivity Index (IRI; Davis, 1983). | Week 0, week 5, and week 10
  The IRI is a self-report measure of empathy, including both cognitive and emotional dimensions. The IRI has 28 items, each rated on a 5-point Likert scale from 0 = does not describe me well to 4 = does describe me very well.

CONTACTS AND LOCATIONS:
Overall Officials: Ole K. Østergård, PhD, Principal Investigator — Department of Communication and Psychology, Aalborg University.; Stig B. Poulsen, Professor, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - Department of Communication and Psychology, Aalborg University, Rendsburggade 14, Aalborg
  - Department of Psychology, University of Copenhagen, Øster Farimagsgade 2A, Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson T, Patterson C. Facilitative Interpersonal Skill Task and Rating Method. Athens: Ohio University; 2013
- [Background] Anderson T, Perlman MR, McCarrick SM, McClintock AS. Modeling therapist responses with structured practice enhances facilitative interpersonal skills. J Clin Psychol. 2020 Apr;76(4):659-675. doi: 10.1002/jclp.22911. Epub 2019 Dec 18. PMID 31851382
- [Background] Lent RW., Hill CE, Hoffman MA. Development and validation of the Counselor Activity Self-Efficacy Scales. Journal of Counseling Psychology. 2003;, 50(1): 97-108. doi: 10.1037//0022-0167.50.1.97.
- [Background] Davis MH. Measuring individual differences in empathy: Evidence for a multidimensional approach. Journal of Personality and Social Psychology. 1983; 44(1): 113-126. doi:10.1037/0022-3514.44.1.113.
- [Background] Benjamin LS. Intrex User's Manual. Salt Lake City: Univ. Utah; 2000.
- [Background] Riggio RE. Manual for the social skills inventory. Palo Alto, CA: Consulting Psychologists Press; 1989
- [Background] Brennan KA, Clark CL, Shaver PR. Self-report measurement of adult attachment: An integrative overview. In: Simpson JA, Rholes WS, editors, Attachment theory and close relationships. New York: Guilford Press; 1998. p. 46-76.
- [Background] Herold DM, Parsons CK, Rensvold RB. Individual differences in the generation and processing of performance feedback. Educational and Psychological Measurement. 1996; 56(1): 5-25. doi:10.1177/0013164496056001001.
- [Background] MacKenzie KR. The clinical application of a Group Climate measure. In: Dies RR, MacKenzie KR, editors. Advances in group psychotherapy: Integrating research and practice. New York: International Universities Press; 1983. p. 159-170.
- [Background] Rousmaniere TG. DP Coach Competency Scale (DPCCS). 2020. Retrieved from https://drive.google.com/file/d/1YySX8avhPaAYm8T4Opvf5QwPwWU0CwLd/view
- [Derived] Ostergard OK, Nielsen J, Hjorthoj C, Nilsson KK, Poulsen SB. Effect of deliberate practice training of graduate students in general psychotherapeutic skills compared with theoretical teaching: protocol for the randomised controlled TRIPS trial. BMJ Open. 2022 Sep 29;12(9):e062506. doi: 10.1136/bmjopen-2022-062506. PMID 36175107